CLINICAL TRIAL: NCT06452160
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of BGC515 Capsules in Patients With Advanced Solid Tumors
Brief Title: A Study of BGC515 Capsules in Subjects With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BridGene Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BGC515-101
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Mesothelioma; Epithelioid Hemangioendothelioma(EHE); Solid Tumor
MeSH Terms: conditions — Mesothelioma; Hemangioendothelioma, Epithelioid

STUDY DESIGN:
Intervention Model Description: Sequential Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): BGC515 Capsules will be administered orally in 21 day cycles, once daily (QD). Patients will be enrolled into escalating dose levels during the Dose Escalation Phase to determine the Maximum Tolerated Dose (MTD) and the Recommended Dose(s) for Expansion (RDE).
  Interventions: Drug: BGC515
- Dose Expansion (Experimental): BGC515 Capsules will be administered orally in 21 day cycles at MTD/RDE defined dose,once daily (QD), in patients with malignant mesothelioma (MM), epithelioid hemangioendothelioma (EHE), or other advanced solid tumors.
  Interventions: Drug: BGC515

INTERVENTIONS:
Drug: BGC515 — Capsules for oral administration

SUMMARY:
The goal of this open-label, dose escalation and dose expansion Phase I clinical trial is to evaluate the safety, tolerability, pharmacokinetics and preliminary efficacy of BGC515 administered once daily in 3 weeks cycles in solid tumor patients.

ELIGIBILITY:
Inclusion Criteria:

* Having signed the written Informed Consent Form
* Male or female aged ≥18 years
* Life expectancy ≥12 weeks
* Eastern Cooperative Oncology Group (ECOG) Performance Score 0 or 1
* Dose escalation phase: Histologically or cytologically confirmed locally advanced or metastatic mesothelioma (MM), epithelioid hemangioendothelioma (EHE), or other advanced solid tumors who have experienced progressive disease or treatment intolerability after receiving the standard-of-care, or refuse to receive or have no access to the standard-of-care
* Dose expansion phase: Histologically or cytologically confirmed locally advanced or metastatic MM, EHE, etc. regardless of Hippo signaling pathway abnormalities, or other advanced solid tumors with Hippo signaling pathway abnormalities, who have experienced progressive disease or treatment intolerability after receiving the standard-of-care, or refuse to receive or have no access to the standard-of-care
* At least one measurable lesion

Exclusion Criteria:

* Previous or current use of transcriptional enhanced associate domain (TEAD) inhibitors
* Inadequate wash-out of prior therapies described per protocol
* Patients with severe or unstable systemic disease, unstable or symptomatic Central Nervous System (CNS) metastasis
* Clinically significant cardiovascular disease as defined in the protocol
* Women who are pregnant or breastfeeding
* Hypersensitivity to the active pharmaceutical ingredient or any excipient of BGC515
* Study staff member or relative of a study staff member directly related to this clinical trial, or a subordinate of the Investigator in this trial or an employee of the Sponsor, though not directly related to this trial
* Serious systemic diseases or laboratory abnormalities or other conditions that, at the Investigator's discretion, will make it unsuitable for the patient to participate in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs). | Through study completion, approximately 1 year.
  AEs will be graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0. AE evaluation will be based on laboratory tests, vital signs, physical examination, and 12-lead electrocardiogram, etc.
Dose-limiting toxicities (DLTs) | Within 24 days after the first dose of study drug.
  DLT refers to the pre-specified AEs that occurred within 24 days after the first dose of study drug.
Objective response rate (ORR) | Through study completion, approximately 3 years.
  Defined as the percentage of participants having complete response (CR) or partial response (PR). Evaluated by the Investigator based on modified Response Evaluation Criteria in Solid Tumors (mRECIST) or Response Evaluation Criteria in Solid Tumors (RECIST) V1.1.
Progress-free survival(PFS) | Through study completion, approximately 3 years.
  Defined as the time interval between the first dose of the treatment and the first documented disease progression or death due to any cause (whichever occurs first). Evaluated by the Investigator based on modified Response Evaluation Criteria in Solid Tumors (mRECIST) or Response Evaluation Criteria in Solid Tumors (RECIST) V1.1.

SECONDARY OUTCOMES:
Peak concentration (Cmax). | Multiple time points, up to approximately 1 year.
  Cmax of BGC515 in plasma.
Time to peak concentration (Tmax). | Multiple time points, up to approximately 1 year.
  Tmax of BGC515 in plasma.
Half-life (t1/2). | Multiple time points, up to approximately 1 year.
  t1/2 of BGC515 in plasma.
Area under the concentration-time curve from time zero to the last detectable plasma concentration (AUC0-t). | Multiple time points, up to approximately 1 year.
  (AUC0-t) of BGC515 in plasma.

CONTACTS AND LOCATIONS:
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No